CLINICAL TRIAL: NCT01569906
Title: Narrowband Ultraviolet B Phototherapy in Children With Moderate to Severe Atopic Eczema- an Observational Prospective Controlled Study
Brief Title: Narrowband UVB for Children With Moderate to Severe Atopic Eczema
Status: Completed | Type: Observational
Sponsor: Royal Victoria Infirmary (Other)
Collaborators: British Skin Foundation (Unknown)
Responsible Party: Principal Investigator, Dr AEM Taylor, Consultant Dermatologist, Royal Victoria Infirmary
Other Study IDs: 4795; 7282 (Other: NIHR)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Moderate to Severe Atopic Eczema
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- UVB: Children with moderate to severe atopic eczema who undertook a standard course of narrowband Ultraviolet B (NBUVB) phototherapy
  Interventions: Radiation: Narrowband Ultraviolet B phototherapy
- Controls: Children with moderate to severe atopic eczema who were offered UVB but were unable to undertake treatment

INTERVENTIONS:
Radiation: Narrowband Ultraviolet B phototherapy — Twice weekly exposures for a total of 24 exposures using a standard phototherapy protocol.
  Groups: UVB

SUMMARY:
To assess prospectively, the response of moderate to severe atopic eczema to a standard course of narrowband ultraviolet B phototherapy by using validated objective and subjective scoring systems.

DETAILED DESCRIPTION:
Children with moderate to severe atopic eczema prescribed a course of narrowband UVB phototherapy were scored (using validated scoring systems) objectively and subjectively before, during and after the course of treatment, as well as 3 and 6 months post treatment (to determine length of remission). Their scores were compared to a control group. The control group comprised children with moderate to severe atopic eczema who were offered UVB but were unable to undertake the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3-16 years with moderate to severe atopic eczema (as defined by the modified Hannifin and Rajka criteria) in whom there is a clinical indication for phototherapy (as deemed by their specialist Dermatology consultant).

Exclusion Criteria:

* Children under the age of 3 years or any child who lacks the maturity needed to stand in the phototherapy cabinet unsupervised.
* Mild disease (defined as a Six Area Six Sign Atopic Dermatitis (SASSAD) score <10)

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3-16 years
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Score at the end of treatment compared to the control group | 12 weeks
  Measurement of Six Area Six Sign Atopic Dermatitis (SASSAD) score and percentage surface area affected of those treated with narrowband UVB as compared to a control group

SECONDARY OUTCOMES:
Subjective scores at the end of treatment as compared to controls | 12 weeks
  Subjective scoring using Patient Outcome Eczema Measure (POEM), Children's Dermatology Life Quality Index (CDLQI), Dermatitis Family Impact Questionnaire (DFI), Visual analogue scale (VAS) for itch and sleep loss
objective scores at 3 months post treatment compared to controls | 3 months
  Objective Six Area Six Sign Atopic Dermatitis (SASSAD) score and percentage surface area affected in the treated group at 3 months post treatment as compared to controls.
Association of filaggrin status with outcome | 12 weeks
  To determine if response to phototherapy is determined by the presence of a homozygous or compound heterozygous filaggrin mutation.
Subjective scores at 3 months post treatment compared to controls | 3 months
  Subjective scores (Patient Outcome Eczema Measure (POEM),Children's Dermatology Life Quality Index (CDLQI), Dermatitis Family Impact Questionnaire (DFI), Visual Analogue Scale (VAS) for itch and sleep loss) in the treated group at 3 months post treatment as compared to controls.
Subjective scores at 6 months post treatment compared to controls | 6 months
  Subjective scores (Patient Outcome Eczema Measure (POEM),Children's Dermatology Life Quality Index (CDLQI), Dermatitis Family Impact Questionnaire (DFI), Visual Analogue Scale (VAS) for itch and sleep loss) in the treated group at 6 months post treatment as compared to controls.
Objective scores at 6 months post treatment compared to controls | 6 months
  Objective Six Area Six Sign Atopic Dermatitis (SASSAD) score and percentage surface area affected in the treated group at 6 months post treatment as compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Aileen EM Taylor, MBChB, Principal Investigator — Royal Victoria Infirmary
Locations (1):
- Royal Victoria Infirmary, Newcastle upon Tyne, United Kingdom